CLINICAL TRIAL: NCT07250399
Title: Effect of Instrumentation Kinematics on Intraoperative and Post-operative Pain in Maxillary Premolars With Acute Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Effect of Instrumentation Kinematics on Intraoperative and Post-operative Pain in Maxillary Premolars With Acute Irreversible Pulpitis
Acronym: Instrumentatio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sabah Morad Sobhy, Endodontic department, al azhar university. principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-PD-25-32
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: the Effect of Instrumentation Kinematics on Intraoperative and Post-operative Pain
Keywords: instrumentation kinematics; post-operative pain; acute irreversible pulpitis
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I reciprocating system (EdgeOne Fire group) (Experimental): Root canal preparation will be completed using EdgeOne Fire reciprocating system (Albuquerque, NM, USA) up to size (35/0.04). Files will be operated at reciprocating motion, where the angle of reciprocation will be set at 150° counterclockwise (CCW) and 30° clockwise (CW).
  Interventions: Device: EdgeOne Fire reciprocating system
- Group II rotary system (JZ file group) (Experimental): Root canal preparation will be completed using JZ file system up to size (35/0.04). The files will be operated at 300 rpm and 2 Ncm torque.
  Interventions: Device: JZ file system

INTERVENTIONS:
Device: EdgeOne Fire reciprocating system — Files will be operated at reciprocating motion, where the angle of reciprocation will be set at 150° counterclockwise (CCW) and 30° clockwise (CW)
  Arms: Group I reciprocating system (EdgeOne Fire group)
Device: JZ file system — The files will be operated at 300 rpm and 2 Ncm torque
  Arms: Group II rotary system (JZ file group)

SUMMARY:
Post-endodontic pain refers to the discomfort experienced following endodontic procedures. The incidence of post-operative pain is reported to be 25-40% regardless of the pulp and periradicular condition. It has been shown that pain prevalence declined from 40% in the first 48 h after treatment to 11% 7 days post-treatment. The mechanisms behind post-endodontic pain are complex and multifactorial that include host-dependent factors such as host immunity and preoperative pain history as well as operator-related factors such as chemical, mechanical or bacterial injury that occurs during endodontic procedure. A major contributor to this pain is the extrusion of infected debris as dentin chips, microorganisms, and the remnants of pulp tissue to the periradicular area. The intensity of pain is directly proportional to the extent of tissue injury caused.

During root canal preparation, a variety of materials including dentin debris, pulp remnants, microorganisms, endotoxins, and irrigating solutions may be extruded into the periapical tissues, potentially leading to inflammation, increased vascular permeability, oedema, nerve compression and postoperative pain. Studies suggest that apical extrusion is affected by file systems, file kinematics and instrumentation techniques used during root canal preparation .

Rotary systems vary in the amount of debris they extrude due to variations in cross-sectional design, flute depth, cutting blade, kinematics, taper, file sequence, tip size and cutting efficiency. Both rotary and reciprocating NiTi files are effective in reducing endotoxins and bacterial by-products from infected root canals. NiTi files enhance biomechanical preparation and canal centering and exhibit greater resistance to cycle fatigue due to their super elasticity and

greater flexibility. However, the extent of periapical inflammation may differ among NiTi systems due to variations in the amounts of extruded irritantsEdgeOne Fire reciprocating system (EdgeEndo, Albuquerque, New Mexico, USA) features a parallelogram cross-section having two cutting edges and an off-center design. these endodontic instruments are treated with a proprietary heat process called FireWire™, that it is claimed to provide high flexibility and a negligible restoring force. It operates using alternating cutting and releasing angles through a reciprocating motion; with an exchange in the direction of rotation.

Jizai rotary file systems (JZ) (MANI, Tochigi, Japan) is a recently developed NiTi rotary system made of a proprietary heat-treated NiTi alloy. JZ system exhibits bending deformation indicating that it is not purely austenitic but contains R-phase and/or martensite at room or body temperature. It has an off-center quasi-rectangular cross-section with a radial land on one of the short sides. According to the manufacturer, this cross-sectional design produces low screw-in forces owing to the radial land and provides wide spaces for debris removal. EdgeOne Fire reciprocating system (EdgeEndo, Albuquerque, New Mexico, USA) features a parallelogram cross-section having two cutting edges and an off-center design. these endodontic instruments are treated with a proprietary heat process called FireWire™, that it is claimed to provide high flexibility and a negligible restoring force. It operates using alternating cutting and releasing angles through a reciprocating motion; with an exchange in the direction of rotation.

Jizai rotary file systems (JZ) (MANI, Tochigi, Japan) is a recently developed NiTi rotary system made of a proprietary heat-treated NiTi alloy. JZ system exhibits bending deformation indicating that it is not purely austenitic but contains R-phase and/or martensite at room or body temperature. It has an off-center quasi-rectangular cross-section with a radial land on one of the short sides. According to the manufacturer, this cross-sectional design produces low screw-in forces owing to the radial land and provides wide spaces for debris removal.A systematic review of the literature suggested that debris extrusion is influenced by instrument kinematics . However, evidence is still conflicting and sometimes even contradicting regarding the association of kinematics with debris extrusion and post-operative pain.

DETAILED DESCRIPTION:
1. Trial design:

   This study will be a parallel randomized controlled trial a. It is written in accordance with the Preferred Reporting Items for Randomized Trial in Endodontics (PRIRATE) 2020 guidelines .
2. Participants:

   Patients of age range between 20 and 50 years old from the outpatient clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University will participate in this study. These patients have maxillary premolar teeth with symptomatic pulpitis. Patients will be informed about all the study's procedures. They will be included in the study after fulfilling the inclusion criteria and sign an informed consent . The Visual Analog Scale (VAS) will be explained to all participants utilizing visual, verbal and numerical methods to ensure complete understanding. Training on its use will be provided after their recruitment and before randomization to ensure that participants are familiar with the scale before pretreatment pain assessment.
3. Sample size calculation:

Sample size calculation was performed using G*Power version 3.1.9.7 based on the results of a previous study (Kherlakian et al.) . A power analysis was designed to have adequate power to apply a two-sided statistical test to reject the null hypothesis that there is no difference between groups. By adopting an alpha level of (0.05) and a beta of (0.2), i.e. power = 80% and an effect size (d) of (0.826). The predicted sample size (n) was (50), i.e., 25 subjects per group. This number is increased to 28 subjects per group to compensate for a drop-out rate of 10%.

Criteria of patient selection:

Inclusion Criteria:

1. Maxillary first and second bi-rooted premolar teeth having type I root canal.
2. Patients have mature teeth with closed apex.
3. Teeth with prolonged response to the pulp tests.
4. Spontaneous pain (preoperative visual analog scale score )4-6).
5. Teeth with normal periapical appearance.
6. Restorable teeth.
7. Patients who will be able to understand the informed consent form and pain recording scales used in the study will be included.

Exclusion Criteria:

1. Patients with apical periodontitis.
2. Patients who received analgesics or anti-inflammatory drugs in the last 12 hours and

   antibiotics for the last 1 month.
3. Presence of multiple teeth that require treatment.
4. Systemic disease.
5. Physical or mental disability.
6. Teeth with calcified root canal, root resorption and tooth mobility.
7. The presence of additional roots or canal variations from maxillary premolar anatomy.
8. Patient unable to tolerate comple¬tion of root canal treatment in a single visit.

Proper diagnosis of the case including patient history, clinical examination, thermal pulp tests and preoperative periapical radiograph will be obtained.

Symptomatic pulpitis will be diagnosed clinically based on positive response to pulp sensibility tests and the presence of spontaneous provoked pain that lasts longer than 30 s. Patients will be asked to record their pretreatment pain level using Visual Analogue Scale (VAS).

Randomization and blinding

Fifty-six patients will be divided randomly into two groups (28 patients in each group) using simple randomization procedure using random number generator. https://www.random.org/ based on the type of file system used.

Both patient and statistician will be blinded to group allocation.

Treatment protocol:

Local anesthesia will be achieved using 2 mL of 4% articaine and 1:100000 epinephrine (Ultracaine DS Fort; Hoechst- Marion Roussel, Frankfurt, Germany). Access cavity will be prepared under strict aseptic condition and rubber dam isolation using diamond round bur and Endo Z bur (Dentsply, Maillfer, Switzerland). The working length will be determined using an electronic apex locator (EAL) and will be confirmed using periapical radiograph. Glide path preparation will be performed manually up to sizes #20K file.

Subsequently, two groups will be formed according to the predetermined group numbers based on the file system to be used in root canal preparation and the operator will be informed with the study group at this phase.

Group I reciprocating system (EdgeOne Fire group):

Root canal preparation will be completed using EdgeOne Fire reciprocating system (Albuquerque, NM, USA) up to size (35/0.04). Files will be operated at reciprocating motion, where the angle of reciprocation will be set at 150° counterclockwise (CCW) and 30° clockwise (CW).

Group II rotary system (JZ file group):

Root canal preparation will be completed using JZ file system up to size (35/0.04). The files will be operated at 300 rpm and 2 Ncm torque.

The files will be operated passively using an endodontic motor Motopex endodontic motor (Woodpecker, Guilian, China). After each file use, the root canal will be irrigated with 5ml of freshly prepared 2.5% sodium hypochlorite (NaOCl) solution (Alex. Deteregents and Chemical Co., Egypt) for 1 minute using a 30-gauge Navi-Tip flexible irrigating needle (Navi-Tip, Ultradent product, South Jourdan, UT). The needle will be inserted into the root canal 2 mm short of the working length without binding. 5 ml of 17% EDTA (Colgate Oral Care Company, Waverly, Australia) for 1 min will be used for smear layer removal following saline separation. 5 ml of saline solution will be used for final irrigation of the root canal to neutralize all the previously used irrigants.

Finally, the root canal system will be obturated using ADSEAL resin-based sealer (Meta Biomed Co, Cheongju, Korea) and gutta-percha (Dentsply Maillefer, Switzerland) with cold lateral condensation method after being completely dried using paper points of comparable size to the master cone. A final coronal restoration with direct composite filling (Filtek Bulk Fill,3M ESPE, USA) will be performed in the same visit.

The patients will be notified about the possible development of pain and given the VAS form to record the pain level. In this scale, the level of pain is specified by using numbers between 0 and 10; no pain (0), mild pain (1-3), moderate pain (4-6) and severe pain (7-10). Ibuprofen 400 mg will be prescribed to patients to be taken only when needed. The VAS scores will be recorded at 6, 12, 24, 48, ,72 h and 1 week as well as analgesic intake.

Intraoperative and postoperative pain and analgesic intake assessment:

* The evaluation of intraoperative pain will be conducted immediately after root canal preparation with each of the instrumentation kinematics using Visual Analog Scale (VAS). In each group, the patients will be asked to specify the level of pain for the buccal and palatal canals separately. The average of two values reported by the patient will be taken and then accepted as VAS value.
* Postoperative pain will be recorded after 6,12,24,48,72 hours and 1 week of the treatment using Visual Analog Scale (VAS).
* Analgesic intake will also be recorded.

Statistical Analysis Data will be collected and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary first and second bi-rooted premolar teeth having type I root canal.
* have mature teeth with closed apex.
* Teeth with prolonged response to the pulp tests.
* Spontaneous pain (preoperative visual analog scale score )4-6).
* Teeth with normal periapical appearance.
* Restorable teeth.
* Patients who will be able to understand the informed consent form and pain recording scales used in the study will be included.

Exclusion Criteria:

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pain | immediately after root canal preparation
  The evaluation of intraoperative pain will be conducted immediately after root canal preparation with each of the instrumentation kinematics using Visual Analog Scale (VAS). In each group, the patients will be asked to specify the level of pain for the buccal and palatal canals separately. The average of two values reported by the patient will be taken and then accepted as VAS value.
Postoperative pain | 6,12,24,48,72 hours and 1 week
  Postoperative pain will be recorded after 6,12,24,48,72 hours and 1 week of the treatment using Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Analgesic intake assessment | from immediately after the treatment to 1 week postoperatively
  Analgesic intake will also be recorded from immediately after the treatment to 1 week postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sabah M Sobhy, PHD, Principal Investigator — Al-Azhar University
Locations (1):
- from the outpatient clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad MZ, Sadaf D, MacBain MM, Merdad KA. Effect of mode of rotation on apical extrusion of debris with four different single-file endodontic instrumentation systems: Systematic review and meta-analysis. Aust Endod J. 2022 Apr;48(1):202-218. doi: 10.1111/aej.12612. Epub 2022 Mar 7. PMID 35255170
- [Background] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285